CLINICAL TRIAL: NCT05583825
Title: The Effect of Rebozo Application in the Intrapartum Period on Labor Pain, Anxiety and Birth Experience
Brief Title: The Effect of Rebozo Application in the Intrapartum Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Zeliha Turan, Principal Investigator, Inonu University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 4463
Record Dates: First submitted 2022-10-04; First posted 2022-10-18 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Birth Order
Keywords: Rebozo App; Birth Pain; Anxiety; Birth Experience
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The status of the participants in the experimental or control group was determined by simple random sampling method. Accordingly, the sample calculation was created by logging into the site https://www.randomizer.org/.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rebozo Applied Group (Experimental): * Those who are in the latent phase (cervical opening 1-4 cm) will be provided to sign the informed consent form by making a statement regarding the research. The Personal Information Form will be filled and the anxiety levels of women with a cervical dilation of 3-4 cm will be determined with the State Anxiety Inventory and the pain level will be determined with the Visual Analog Scale, and rebozo techniques will be applied two or three times. After the application, the level of pain will be re-evaluated.
  * When the cervical dilation is 6-7 cm (active phase), the pain level will be determined with the Visual Analog Scale, Rebozo Techniques will be applied two or three times and the pain level will be re-evaluated after the application.
  * When the cervical opening is 8-9 cm (transition phase), the pain level will be determined, Rebozo Techniques will be applied two or three times, and anxiety and pain levels will be evaluated after the application.
  Interventions: Other: Rebozo App
- Standard Care Group (No Intervention): * Pregnant women who will not be subjected to any application other than routine hospital applications, who are in the latent phase (cervical opening 1-4 cm), will be provided to sign the informed consent form by making a statement about the research. Afterwards, by filling out the Personal Information Form, the anxiety levels of women with a cervical dilation of 3-4 cm will be determined with the State Anxiety Inventory, and their pain levels will be determined with the Visual Analog Scale.
  * When the cervical opening is 6-7 cm (active phase), the level of pain will be determined.
  * When the cervical dilation is 8-9 cm (transition phase), anxiety and pain levels will be determined.
  * The Travay Follow-up Form will be used in the period from the admission of women to labor until the end of the action.
  * Evaluation of birth experience will be done in the fourth stage of labor using the birth experience scale.

INTERVENTIONS:
Other: Rebozo App — It is a non-invasive, non-drug practical application made with Rebozo, a long and colorful fabric, two meters long and 70 cm wide, worn by Mexican women on their head and shoulders.
  Arms: Rebozo Applied Group

SUMMARY:
This research, which was planned as a randomized experimental control study with intervention to determine the effect of Rebozo application applied to primiparous women during labor, on labor pain, anxiety and birth experience, will be conducted in the Birth Hall of Şanlıurfa Training and Research Hospital. The universe of the research consists of pregnant women who were admitted to the Delivery Hall to perform the labor, and the sample will be a minimum of 62 pregnant women, 31 in the experimental group and 31 in the control group. Research data will be collected by face-to-face interview method using Personal Information Form, Tramway Follow-up Form, Visual Analog Scale (VAS), Spielberger State Anxiety Inventory and Birth Experience Scale. From the pregnant women who met the sampling criteria to the women included in the intervention group; Rebozo techniques will be applied two or three times in each phase (latent phase, active phase and transitional phase), and pregnant women in the control group will not be subjected to any application other than routine hospital applications.

SPSS 24.0 package program will be used in the analysis of the data, and it will be evaluated with descriptive analyzes and correlation analyzes.

With the findings to be obtained as a result of the study, the effect of Rebozo applied to primiparous women during labor on labor pain, anxiety and birth experience will be determined. In addition, scientific evidence for the application of Rebozo will be provided with the data to be obtained.

DETAILED DESCRIPTION:
Birth is one of the most important life experiences of a woman throughout her life. perceived pain at birth; it is a subjective condition that has different feelings for each woman and is affected by physiological, psychological, cultural and environmental factors. In addition to being a physiological indicator of the progress of labor, labor pain, which is multidimensional, can adversely affect maternal and fetal health if an effective pain management is not applied. Therefore, the American Society of Obstetrics and Gynecology (ACOG) recommends appropriate interventions to alleviate labor pain. The application of non-pharmacological methods in the management of pain allows women to see birth as a natural event, but it can be effective in reducing cesarean rates by increasing the satisfaction of the pregnant woman in normal vaginal delivery. In addition, supportive applications in the intrapartum period; It is known to be effective on shortening the birth period, positive outcomes for mothers and newborns, and positive birth and care experiences.

Among the non-pharmacological applications, one of the traditional applications, the Latin American origin, non-invasive Rebozo Technique is located. Rebozo is a long and colorful fabric, two meters long and 70 cm wide, worn by Mexican women on their head and shoulders. Rebozo application is to relieve pain by creating a rhythmic movement in the mother's pelvis and to help the fetus enter a suitable position for delivery by relaxing the pelvic muscles. In addition to relieving pain; It can be applied to many parts of the body because it is effective in times such as low back pain, stress, fatigue, the need for a position change in the baby's womb. This technique is used by midwives or nurses in various positions while the woman is lying down, standing, or on her hands and knees in childbirth. In addition, it can be applied between 5-10 minutes during contractions, or this time can be extended or shortened according to the woman's preference.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years ,
* Able to communicate
* Having a single-vertex and healthy fetus at term,
* No disability or disease,
* Primiparous women who agreed to participate in the study.

Exclusion Criteria:

* Those who are administered sedative and pharmacological drugs during the action process,
* Those who develop maternal or fetal complications,
* Those who received cesarean section for any reason,
* Those who want to leave the research.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Visual Analog Skala (VAS) | In order to determine the effect of rebose on pain, the pain level of women before and after reboza will be evaluated in each phase. Thus, "the change in pain level in approximately 7-10 minutes" will be evaluated in each phase.
  Visual analog scale is a measurement tool used to convert some values that cannot be measured numerically to digital. It measures the severity of pain in individuals. It is a 10 cm long ruler with the phrase "no pain" on the left end and the phrase "unbearable pain" on the right end.As the VAS value approaches 10, the pain is considered to be very severe, and as it approaches 0, the pain decreases.
Spielberger State Anxiety Inventory | To determine the effect of rebozo on state anxiety, the change in women's state anxiety level "(change within approximately 12-14 hours)" will be evaluated just before rebozo in the latent period and immediately after rebozo administration in tr.
  The scale is used to reveal the anxiety experienced by the person at that moment. It is a self-evaluation type scale consisting of short statements. It consists of 20 items.The total score obtained from the scale varies between 20-80. A large score indicates a high level of anxiety, and a small score indicates a low level of anxiety. It is a four-degree scale ranging from "Not at all" to "Totally".
Birth Experience Scale-CEQ | Both the rebozo group and the standard care group; It will be filled in the fourth stage of labor (within the first 4 hours after the delivery of the placenta).
  The purpose of the scale; to evaluate women's birth experiences in different contexts. The scale consists of four sub-dimensions including birth process, professional help/support, perceived security, participation in decisions and 22 items. The first 19 items in the scale are evaluated using a four-point Likert scale and the last three items are evaluated using the Visual Analogue Scale (VAS). The first 19 items are used by scoring from 1 to 4. Scoring is defined as: Totally agree = 1, Mostly agree = 2, Partially agree =3, Strongly disagree = 4. Since the 3rd, 5th, 8th, 9th and 20th items of the scale include negative statements, these items are scored reversed. As the score obtained from the scale increases, it is concluded that the woman has a positive birth experience.

OTHER OUTCOMES:
Personal Information Form (Socio-demographic, obstetric characteristics and thoughts on the method) | At the beginning of the study (in the latent phase), the socio-demographic and obstetric characteristics of women in both the Rebozo group and the standard care group will be evaluated. Then, women who received rebozo in the fourth stage of labor (within
  This form, which was developed by the researcher in line with the literature, consists of five questions containing the socio-demographic characteristics of the women participating in the research (age, education level, employment status, income status, place of residence); five questions including obstetric characteristics (week of pregnancy, planned pregnancy, preparation for birth and training to cope with labor and fear of the birth process); and how the woman evaluates the Rebozo application (the effectiveness of the application on pain, fear/anxiety, whether the application is repeated and recommended, the problems experienced during the application), a total of 15 questions.
Travay Follow-up Form | At the beginning of the study, sections where maternal and fetal findings can be recorded will be filled for women in both groups. All evaluations will continue to be recorded on the form during the period until the birth (average 12-14 hours).
  This form, which was developed by the researcher on the basis of the Partograph Form, was prepared in order to follow the process from the admission of the participants in the study to the delivery. Vaginal examination findings according to the stages of labor, fetal heart rate, contraction characteristics, dose and time of the drugs used, time of birth, duration of the second stage, episiotomy and laceration status, gender, height and weight of the newborn, and APGAR scores at 1 and 5 minutes. place is given.

CONTACTS AND LOCATIONS:
Overall Officials: Yurdagül Yağmur, PhD, Study Chair — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)

REFERENCES:
- [Result] Iversen ML, Midtgaard J, Ekelin M, Hegaard HK. Danish women's experiences of the rebozo technique during labour: A qualitative explorative study. Sex Reprod Healthc. 2017 Mar;11:79-85. doi: 10.1016/j.srhc.2016.10.005. Epub 2016 Oct 31. PMID 28159133
- [Derived] Turan Z, Yagmur Y. The Effect of Rebozo Massage on Birth Pain, Anxiety, and Childbirth Experience in the Intrapartum Period: A Randomized Controlled Trial in Turkiye. J Transcult Nurs. 2026 Jan;37(1):137-147. doi: 10.1177/10436596251366932. Epub 2025 Sep 12. PMID 40936453